CLINICAL TRIAL: NCT02823470
Title: A Phase 4, Open-label Treatment, Randomized, Multicenter, 2-arm, Parallel-group, Pilot Study of Adherence to Lumacaftor/Ivacaftor in CF Subjects Homozygous for the F508del CFTR Mutation
Brief Title: A Pilot Study to Evaluate the Use of Smart Adherence Technology to Measure Lumacaftor/Ivacaftor Adherence in CF Subjects Homozygous for the F508del CFTR Mutation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated early due to slow recruitment of patients.
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VX15-809-114
Record Dates: First submitted 2016-07-01; First posted 2016-07-06 (Estimated); Results first posted 2018-09-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-08

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — lumacaftor, ivacaftor drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: activated smart device alerts and feedback (Experimental): LUM/IVA: LUM 400 mg q12h/IVA 250 mg q12h through Week 48.
  Interventions: Drug: LUM/IVA; Device: activated smart device
- Arm B: de-activated smart device alerts/feedback features (Experimental): LUM/IVA: LUM 400 mg q12h/IVA 250 mg q12h through Week 48.
  Interventions: Drug: LUM/IVA; Device: de-activated smart device

INTERVENTIONS:
Drug: LUM/IVA — LUM 400 mg q12h/IVA 250 mg q12h through Week 48.
  Other Names: lumacaftor/ivacaftor
Device: activated smart device
  Arms: Arm A: activated smart device alerts and feedback
Device: de-activated smart device
  Arms: Arm B: de-activated smart device alerts/feedback features

SUMMARY:
The study will evaluate the impact of smart adherence technology for monitoring on lumacaftor/ivacaftor (LUM/IVA) adherence rates among subjects 16 years of age and older with Cystic Fibrosis (CF) who are homozygous for the F508del Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) mutation.

ELIGIBILITY:
Inclusion Criteria:

* Subject (or his or her legally appointed and authorized representative) will sign and date an informed consent form (ICF).
* Willing and able to comply with scheduled visits, treatment plan, study restrictions, laboratory tests, contraceptive guidelines, and other study procedures.
* Confirmed diagnosis of CF and homozygous for the F508del-CFTR mutation
* Forced Expiratory Volume in one second/forced vital capacity (FEV1) ≥40% of predicted normal for age, sex, and height

Exclusion Criteria:

* Presence of moderate or severe hepatic impairment (Child-Pugh Class B or C)
* Subjects currently receiving invasive mechanical ventilation
* Known history of alcohol or drug abuse in the past year
* Clinically significant abnormal laboratory values during screening
* Pregnant or nursing females
* Female subjects and female partners of male subjects who plan to become pregnant during Treatment Period or within 90 days following the last dose of study drug
* History of solid organ or hematological transplantation
* Ongoing or prior participation in an investigational drug study within 30 days of screening
* Current use of commercial LUM/IVA combination therapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-06; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (7):
  - Hartford, Connecticut
  - Washington D.C., District of Columbia
  - Orlando, Florida
  - Atlanta, Georgia
  - Jackson, Mississippi
  - Albuquerque, New Mexico
  - Columbia, South Carolina
- Canada (4):
  - Edmonton, Alberta
  - Victoria, British Columbia
  - Saint John, New Brunswick
  - Québec

RESULTS

PARTICIPANT FLOW:
Groups:
- LUM/IVA Through Deactivated Smart Pill Bottle (Control): Participants received lumacaftor (LUM) 400 milligram (mg) in combination with ivacaftor (IVA) 250 mg as oral tablet every 12 hours (q12h) for up to 35 weeks through a de-activated smart pill bottle (control).
- LUM/IVA Through Activated Smart Pill Bottle (Test): Participants received LUM 400 mg in combination with IVA 250 mg as oral tablet q12h for up to 35 weeks through an activated smart pill bottle.
Period: Overall Study
Arm/Group | LUM/IVA Through Deactivated Smart Pill Bottle (Control) | LUM/IVA Through Activated Smart Pill Bottle (Test)
Started | 9 | 15
Completed | 0 | 0
Not Completed | 9 | 15
Not completed — Adverse Event | 1 | 0
Not completed — Study terminated by sponsor | 8 | 15

BASELINE CHARACTERISTICS:
Groups:
- LUM/IVA Through Deactivated Smart Pill Bottle (Control): Participants received LUM 400 mg in combination with IVA 250 mg as oral tablet q12h for up to 35 weeks through a de-activated smart pill bottle (control).
- Total: Total of all reporting groups
Arm/Group | LUM/IVA Through Deactivated Smart Pill Bottle (Control) | LUM/IVA Through Activated Smart Pill Bottle (Test) | Total
Number analyzed (Participants) | 9 | 15 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 20.8 (4.0) | 25.1 (10.3) | 23.5 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 4 | 9 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 15 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 15 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage Adherence to Lumacaftor/Ivacaftor (LUM/IVA) Treatment
Description: Percentage adherence was reported in terms of median and full range due to small sample size.
Time Frame: Up to 35 weeks
Population: Full analysis set (FAS) included randomized participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: percentage of adherence
Arm/Group | LUM/IVA Through Deactivated Smart Pill Bottle (Control) | LUM/IVA Through Activated Smart Pill Bottle (Test)
Number analyzed (Participants) | 9 | 15
percentage of adherence | 85.49 [32.0 to 96.4] | 92.07 [74.2 to 99.3]

2. Secondary Outcome: Percentage Adherence to Lumacaftor/Ivacaftor (LUM/IVA) Treatment Through 12 Weeks
Description: Percentage adherence was reported in terms of median and full range due to small sample size.
Time Frame: Up to Week 12
Population: FAS included randomized participants who received at least 1 dose of study drug. "Overall Number of Participants Analyzed" signifies those participants who had at least 12 weeks of eligible smart pill bottle data.
Measure: Median (Full Range); unit: percentage of adherence
Arm/Group | LUM/IVA Through Deactivated Smart Pill Bottle (Control) | LUM/IVA Through Activated Smart Pill Bottle (Test)
Number analyzed (Participants) | 6 | 14
percentage of adherence | 88.69 [37.5 to 94.0] | 97.32 [74.4 to 100.0]

3. Secondary Outcome: Number of Participants With Greater Than or Equal to (>=) 80 Percent (%) Adherence
Description: Number of participants with >=80% adherence to LUM/IVA treatment over 12 weeks were reported.
Time Frame: Up to Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- LUM/IVA Through Deactivated Smart Pill Bottle (Control): Participants received lumacaftor (LUM) 400 milligram (mg) in combination with ivacaftor (IVA) 250 mg as oral tablet every 12 hours (q12h) for up to 35 weeks through a de-activated smart pill bottle.
- LUM/IVA Through Activated Smart Pill Bottle (Test): Participants received lumacaftor (LUM) 400 milligram (mg) in combination with ivacaftor (IVA) 250 mg as oral tablet every 12 hours (q12h) for up to 35 weeks through an activated smart pill bottle.
Arm/Group | LUM/IVA Through Deactivated Smart Pill Bottle (Control) | LUM/IVA Through Activated Smart Pill Bottle (Test)
Number analyzed (Participants) | 6 | 14
Participants | 4 | 13

4. Secondary Outcome: Number of Participants With Greater Than or Equal to (>=) 90 Percent (%) Adherence
Description: Number of participants with >=90% adherence to LUM/IVA treatment over 12 weeks were reported.
Time Frame: Up to Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- LUM/IVA Through Deactivated Smart Pill Bottle (Control): Participants received LUM 400 mg in combination with IVA 250 mg as oral tablet q12h for up to 35 weeks through a de-activated smart pill bottle.
Arm/Group | LUM/IVA Through Deactivated Smart Pill Bottle (Control) | LUM/IVA Through Activated Smart Pill Bottle (Test)
Number analyzed (Participants) | 6 | 14
Participants | 2 | 12

ADVERSE EVENTS:
Time Frame: Baseline up to Week 35
Arm/Group | LUM/IVA Through Deactivated Smart Pill Bottle (Control) | LUM/IVA Through Activated Smart Pill Bottle (Test)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/15
Other Adverse Events (participants affected / at risk) | 4/9 | 9/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LUM/IVA Through Deactivated Smart Pill Bottle (Control) (N=9) | LUM/IVA Through Activated Smart Pill Bottle (Test) (N=15)
Cholecystitis (Hepatobiliary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LUM/IVA Through Deactivated Smart Pill Bottle (Control) (N=9) | LUM/IVA Through Activated Smart Pill Bottle (Test) (N=15)
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 3
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 1 | 0
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Headache (Nervous system disorders) | 0 | 2
Loss of consciousness (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Cystic fibrosis related diabetes (Congenital, familial and genetic disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
As a result of the early termination, definitive conclusions cannot be made given the limited sample size and incomplete data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is free to publish results of the study after (1) the first multi-center publication, (2) if the sponsor elects not to publish the results, or (3) 18 months after close of the study, whichever occurs first. Proposed publications are to be submitted to the sponsor for review and comment for a period of at least 45 days (which may be extended under certain circumstances related to protection of intellectual property); the sponsor cannot require changes to the proposed publications.

DOCUMENTS (2):
  • Study Protocol (2016-10-19): https://cdn.clinicaltrials.gov/large-docs/70/NCT02823470/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-15): https://cdn.clinicaltrials.gov/large-docs/70/NCT02823470/SAP_001.pdf